CLINICAL TRIAL: NCT03034200
Title: Phase 2 Study of ONC201 in Neuroendocrine Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peter Anderson (Other)
Responsible Party: Sponsor-Investigator, Peter Anderson, Site Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE2716
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Recurrent Neuroendocrine Tumor; Metastatic Neuroendocrine Tumor
Keywords: Pheochromocytoma-paraganglioma; ONC201
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — TIC10 compound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A: Metastatic PC-PG (Experimental): 625mg ONC201 will be given once weekly
  Interventions: Drug: ONC201
- Arm B: Other NETs (Experimental): 625mg ONC201 will be given once weekly
  Interventions: Drug: ONC201
- Arm C: PC-PG + other NETs (Experimental): 625mg ONC201 will be given on day 1 and day 2 of each week
  Interventions: Drug: ONC201

INTERVENTIONS:
Drug: ONC201 — 625mg ONC201 will be given on two consecutive days each week

SUMMARY:
The purpose of this study is to learn if a new drug, ONC201 can make tumors become smaller or go away completely. Investigators also want to learn if ONC201 can prevent new deposits of cancer from appearing in new places in participants (metastases). A phase 2 study of ONC201 in PC-PG (pheochromocytoma-paraganglioma) and other neuroendocrine tumors will determine whether inhibition of DRD2 (a member of the dopamine receptor family) is safe in unresectable, recurrent, locally advanced, refractory, or metastatic neuroendocrine cancers including PC-PG, desmoplastic small round cell tumor (DSRCT), Ewing sarcoma (PNET) or any other neuroendicrine tumor with a catecholamine or dopamine biomarker or autocrine or paracrine dependence on dopamine including cholangiocarcinoma and adrenal cortical carcinoma.

ONC201 is an investigational (experimental) agent and has a favorable safety profile in phase 1 and early phase 2 clinical trials in advanced cancers. This study design has been chosen to see whether ONC201 is associated with reduction of anti-hypertension medications, safety and significant efficacy against neuroendocrine tumors, especially PC-PG.

DETAILED DESCRIPTION:
Primary Objective To demonstrate objective responses using MRI or CT, and/or PET-CT imaging. The same CT or MRI imaging to assess disease burden at study entry will be compared at week 6 and 3 months. Patients without progression at 3 months will continue treatment and have imaging at 6, 9 and 12 months after study entry. Metabolic response and/or biomarkers will be compared with study entry PET-CT and scans at 6 weeks, 3 months and 12 months.

Secondary Objectives Progression - free Survival: This will be calculated according to Response Evaluation Criteria In Solid Tumors (RECIST) or development of new disease

Overall survival: Overall survival will be determined by email or telephone contact.

Study Design: Phase 2 open-label fixed dose study Metastatic neuroendocrine tumors including PC-PG are rare diseases.

The current recommended phase II dose of 625 mg orally on 2 consecutive days every week will be used. The same imaging at study entry will be used at subsequent time points (CT or MRI for week 6 and 3, 6, 9, and 12 months) Imaging modality choice will be influenced by the quality of prior scans of the subject and will be ordered so clinical comparison is possible.

Because of travel and lodging considerations associated with the COVID-19 pandemic, some information by the study team/PI may be obtained using virtual visits and 2nd read of scans sent to Cleveland Clinic

ELIGIBILITY:
1. "Subjects must have a unresectable, recurrent, locally advanced, refractory, or metastatic neuroendocrine tumor including pheochromocytoma-paraganglioma (PC-PG), DSRCT, Ewing Sarcoma or PNET, or any neuroendocrine tumor with a catecholamine or dopamine biomarker or autocrine or paracrine dependence on dopamine including cholangiocarcinoma and adrenal cortical carcinoma (ACC).
2. There is no limit on number of prior therapies.
3. Age ≥14 years.
4. Subjects must have normal organ and marrow function as defined below. Studies should be done within 3 weeks prior to enrollment

   * Hemoglobin ≥ 10.0 g/dl
   * Leukocytes ≥ 1500/mcL
   * Absolute neutrophil count ≥ 1,000/mcL
   * Platelet count ≥ 75000/mcL
   * Total bilirubin within 1.5 x normal institutional limits
   * AST (SGOT) ≤ 5 X institutional upper limit of normal
   * ALT (SGPT) ≤ 5 X institutional upper limit of normal
   * Serum Creatinine <3.0mg/dL

     * 5 1 lesion detectable on CT, MRI, 18FDG PET-CT

6 Subjects must have the ability to understand and the willingness to sign a written informed consent document.

7: Karnofsky or if <16 years old Lansky Play Performance status ≥ 60%

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Anderson, MD, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center
Locations (1):
- Cleveland Clinic Pediatric and Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen JE, Krigsfeld G, Mayes PA, Patel L, Dicker DT, Patel AS, Dolloff NG, Messaris E, Scata KA, Wang W, Zhou JY, Wu GS, El-Deiry WS. Dual inactivation of Akt and ERK by TIC10 signals Foxo3a nuclear translocation, TRAIL gene induction, and potent antitumor effects. Sci Transl Med. 2013 Feb 6;5(171):171ra17. doi: 10.1126/scitranslmed.3004828. PMID 23390247
- [Background] Allen JE, Krigsfeld G, Patel L, Mayes PA, Dicker DT, Wu GS, El-Deiry WS. Identification of TRAIL-inducing compounds highlights small molecule ONC201/TIC10 as a unique anti-cancer agent that activates the TRAIL pathway. Mol Cancer. 2015 May 1;14:99. doi: 10.1186/s12943-015-0346-9. PMID 25927855
- [Background] Allen JE, Prabhu VV, Talekar M, van den Heuvel AP, Lim B, Dicker DT, Fritz JL, Beck A, El-Deiry WS. Genetic and Pharmacological Screens Converge in Identifying FLIP, BCL2, and IAP Proteins as Key Regulators of Sensitivity to the TRAIL-Inducing Anticancer Agent ONC201/TIC10. Cancer Res. 2015 Apr 15;75(8):1668-74. doi: 10.1158/0008-5472.CAN-14-2356. Epub 2015 Feb 13. PMID 25681273
- [Background] Allen JE, Kline CL, Prabhu VV, Wagner J, Ishizawa J, Madhukar N, Lev A, Baumeister M, Zhou L, Lulla A, Stogniew M, Schalop L, Benes C, Kaufman HL, Pottorf RS, Nallaganchu BR, Olson GL, Al-Mulla F, Duvic M, Wu GS, Dicker DT, Talekar MK, Lim B, Elemento O, Oster W, Bertino J, Flaherty K, Wang ML, Borthakur G, Andreeff M, Stein M, El-Deiry WS. Discovery and clinical introduction of first-in-class imipridone ONC201. Oncotarget. 2016 Nov 8;7(45):74380-74392. doi: 10.18632/oncotarget.11814. PMID 27602582
- [Background] Hayes-Jordan AA, Ma X, Menegaz BA, Lamhamedi-Cherradi SE, Kingsley CV, Benson JA, Camacho PE, Ludwig JA, Lockworth CR, Garcia GE, Craig SL. Efficacy of ONC201 in Desmoplastic Small Round Cell Tumor. Neoplasia. 2018 May;20(5):524-532. doi: 10.1016/j.neo.2018.02.006. Epub 2018 Apr 5. PMID 29626752
- [Background] Prabhu VV, Lulla AR, Madhukar NS, Ralff MD, Zhao D, Kline CLB, Van den Heuvel APJ, Lev A, Garnett MJ, McDermott U, Benes CH, Batchelor TT, Chi AS, Elemento O, Allen JE, El-Deiry WS. Cancer stem cell-related gene expression as a potential biomarker of response for first-in-class imipridone ONC201 in solid tumors. PLoS One. 2017 Aug 2;12(8):e0180541. doi: 10.1371/journal.pone.0180541. eCollection 2017. PMID 28767654
- [Background] Anderson PM, Hanna R. Defining Moments: Making Time for Virtual Visits and Catalyzing Better Cancer Care. Health Commun. 2020 May;35(6):787-791. doi: 10.1080/10410236.2019.1587695. Epub 2019 Mar 24. PMID 30907145
- [Result] Anderson PM, Trucco MM, Tarapore RS, Zahler S, Thomas S, Gortz J, Mian O, Stoignew M, Prabhu V, Morrow S, Allen JE. Phase II Study of ONC201 in Neuroendocrine Tumors including Pheochromocytoma-Paraganglioma and Desmoplastic Small Round Cell Tumor. Clin Cancer Res. 2022 May 2;28(9):1773-1782. doi: 10.1158/1078-0432.CCR-21-4030. PMID 35022321

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm B: Other NETs: 625mg ONC201will be given once weekly
Period: Overall Study
Arm/Group | Arm A: Metastatic PC-PG | Arm B: Other NETs | Arm C: PC-PG + Other NETs
Started | 10 | 12 | 8
Completed | 0 | 1 | 0
Not Completed | 10 | 11 | 8
Not completed — Disease progression | 8 | 10 | 4
Not completed — Physician Decision | 2 | 0 | 3
Not completed — Patient off treatment for other complicating disease | 0 | 1 | 0
Not completed — Adjuvant Therapy | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Metastatic PC-PG | Arm B: Other NETs | Arm C: PC-PG + Other NETs | Total
Number analyzed (Participants) | 10 | 12 | 8 | 30
Age, Customized [Count of Participants; unit: Participants] — Age, categorized by age range
  Participants
    0-9 years of age | 0 | 1 | 0 | 1
    10-19 years of age | 1 | 1 | 0 | 2
    20-29 years of age | 0 | 4 | 1 | 5
    30-39 years of age | 2 | 3 | 2 | 7
    40-49 years of age | 2 | 2 | 0 | 4
    50-59 years of age | 2 | 0 | 3 | 5
    60-69 years of age | 2 | 1 | 2 | 5
    70-79 years of age | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 7
  Male | 8 | 9 | 6 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 0 | 1
  Not Hispanic or Latino | 9 | 11 | 8 | 28
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 8 | 11 | 8 | 27
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 10 | 12 | 8 | 30

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response According to RECIST Criteria
Description: Complete Response (CR) Disappearance or fibrosis of all target lesions. Any pathologic lymph nodes must have reduction in short axis to <10mm and standardized uptake value (SUV) is <4.
  Partial Response (PR) At least 30% decrease in sum of longest diameters of target lesions (compared to initial on study baseline) and any decrease in SUV in Fludeoxyglucose 18F (18FDG) imaging Stable disease (SD) 0-29% decrease in sum of longest diameters of target lesions (compared to initial on study baseline) or 0-19% increase in sum of longest diameters of target lesions (compared to initial on study baseline). SUV may increase or decrease Progressive disease 20% or more increase of sum of longest diameters of target lesions (compared to initial on study baseline). The sum must also be at an increase of at least 5mm or one or more new lesions that are considered metastatic disease
Time Frame: Up to 1 Year
Population: All participants were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Metastatic PC-PG | Arm B: Other NETs | Arm C: PC-PG + Other NETs
Number analyzed (Participants) | 10 | 12 | 8
Participants
  Complete Response (CR) | 0 | 0 | 0
  Partial Response (PR) | 5 | 1 | 1
  Stable Disease (SD) | 2 | 2 | 7
  Progressive disease | 3 | 9 | 0

2. Secondary Outcome: Median Duration of Therapy
Description: The median Duration of therapy was measured. Participants with stable disease + PR allowed to continue; participants with progression were taken off therapy.
Time Frame: Up to 5 years
Population: All participants were analyzed for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A: Metastatic PC-PG | Arm B: Other NETs | Arm C: PC-PG + Other NETs
Number analyzed (Participants) | 10 | 12 | 8
months | 9 [1.5 to 33] | 3 [1.5 to 33] | 10 [6 to 21]

3. Secondary Outcome: Overall Survival
Description: Time from beginning of treatment until death, or one year, whichever comes first.
Time Frame: Up to 1 Year
Population: All participants were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Metastatic PC-PG | Arm B: Other NETs | Arm C: PC-PG + Other NETs
Number analyzed (Participants) | 10 | 12 | 8
Participants | 4 | 4 | 7

4. Post Hoc Outcome: Number of Participants With Decline in Karnofsky Performance Status
Description: Participant performance status was measured using Karnofsky Performance Status Scale with the goal of determining the number of participants with a decline in score at 12 weeks. Karnofsky Performance Scale Index is an assessment tool for functional impairment. Scores can range from 0 to 100, with 100 indicating normal performance with no complaints or evidence of disease, while 0 indicates death.
Time Frame: 3 months
Population: All participants were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Metastatic PC-PG | Arm B: Other NETs | Arm C: PC-PG + Other NETs
Number analyzed (Participants) | 10 | 12 | 8
Participants | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Arm A: Metastatic PC-PG | Arm B: Other NETs | Arm C: PC-PG + Other NETs
All-Cause Mortality (participants affected / at risk) | 6/10 | 8/12 | 2/8
Serious Adverse Events (participants affected / at risk) | 3/10 | 1/12 | 4/8
Other Adverse Events (participants affected / at risk) | 4/10 | 1/12 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Metastatic PC-PG (N=10) | Arm B: Other NETs (N=12) | Arm C: PC-PG + Other NETs (N=8)
Cardiac disorders - Other, specify: Abnormal EKG (Cardiac disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Pain (General disorders) | 3 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Infections and infestations - Other, specify: Gram positive infection (Infections and infestations) | 0 | 0 | 2
Nervous system disorders - Other, specify: Spinal cord compression (Nervous system disorders) | 0 | 0 | 1
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hepatic hemorrhage (Hepatobiliary disorders) | 0 | 1 | 0
Thromboembolic event (Vascular disorders) | 0 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Edema face (General disorders) | 1 | 0 | 0
Fever (General disorders) | 1 | 0 | 1
General disorders and administration site conditions - Other, specify - Hives (General disorders) | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Vascular disorders - Other, specify - Hemoptysis (Vascular disorders) | 0 | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Atrial Flutter (Cardiac disorders) | 0 | 0 | 1
Surgical and medical procedures - Other, specify - High volume of bleeding (Surgical and medical procedures) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory, thoracic and mediastinal disorders - Other, specify - Mechanical vent support (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
White blood cell decreased (Investigations) | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Alkalosis (Metabolism and nutrition disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Death NOS (General disorders) | 0 | 0 | 1
Surgical and medical procedures - Other, specify - Exploratory laparotomy of abdomen (Surgical and medical procedures) | 1 | 0 | 0
Serum sickness (Immune system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Metastatic PC-PG (N=10) | Arm B: Other NETs (N=12) | Arm C: PC-PG + Other NETs (N=8)
Spasticity (Nervous system disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Alkaline phosphatase increased (Investigations) | 1 | 0 | 1
Anemia (Blood and lymphatic system disorders) | 2 | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 0 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrial Flutter (Cardiac disorders) | 1 | 0 | 0
Bloating (Gastrointestinal disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Brachial plexopathy (Nervous system disorders) | 1 | 0 | 0
Cardiac disorders - Other, specify: Myopericarditis (Cardiac disorders) | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 1
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0
Confusion (Psychiatric disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Creatinine increased (Investigations) | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 3
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1
Dry Eye (Eye disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Ear and labyrinth disorders - Other, specify: Eustachian tube dysfunctin (Ear and labyrinth disorders) | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1
Fatigue (General disorders) | 2 | 0 | 2
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Fever (General disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal disorders - Other, specify: Neurogenic bowel (Gastrointestinal disorders) | 0 | 0 | 1
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 0 | 1
General disorders and administration site conditions - Other, specify: Facial swelling (General disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other, specify: Hives (General disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other, specify: Neck swelling (General disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 2
Hot flashes (Vascular disorders) | 1 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 3 | 0 | 5
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypertension (Vascular disorders) | 1 | 0 | 4
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 2 | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 3
Investigations - Other, specify: Alkaline phosphatase decreased (Investigations) | 0 | 0 | 1
Investigations - Other, specify: Aspartate aminotransferase decreased (Investigations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1
Metabolism and nutrition disorders - Other, specify: Hyperphosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Metabolism and nutrition disorders - Other, specify: Tube feed (Metabolism and nutrition disorders) | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 3
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1
Pain (General disorders) | 3 | 0 | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 1
Platelet count decreased (Investigations) | 1 | 0 | 2
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Proctitis (Gastrointestinal disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Psychiatric disorders - Other, specify: Dysthymia (Psychiatric disorders) | 0 | 0 | 1
Renal and urinary disorders - Other, specify: Orthotopic bladder (neobladder) (Renal and urinary disorders) | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 1
Skin and subcutaneous tissue disorders - Other, specify: Contact dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Urinary Incontinence (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Vascular disorders - Other, specify: Diaphoresis (Vascular disorders) | 1 | 0 | 0
Ventricular Tachycardia (Cardiac disorders) | 0 | 0 | 1
White blood cell decreased (Investigations) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03034200/Prot_SAP_000.pdf
  • Informed Consent Form (2021-06-30): https://cdn.clinicaltrials.gov/large-docs/00/NCT03034200/ICF_001.pdf